CLINICAL TRIAL: NCT03331055
Title: Percutaneous Electrical Nerve Stimulation or Transcutaneous Electrical Nerve Stimulation for Pain in Patients With Pancreatic Cancer
Brief Title: PENS or TENS for Pain in Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-TCM-01
Record Dates: First submitted 2017-10-28; First posted 2017-11-06 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2018-10

CONDITIONS: Pain; Cancer Pain; Pancreatic Cancer
Keywords: percutaneous electrical nerve stimulation; transcutaneous electrical nerve stimulation; pain; pancreatic cancer
MeSH Terms: conditions — Pain; Cancer Pain; Pancreatic Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: patients with pancreatic cancer pain
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant is allocated randomly by staff A, and grouping situation is concealed; Technician (stuff B) or chargeing docotor operates PENS or TENS, or administers oral analgesic medication; Related datas are collected according to perdetermined forms by stuff C; Outcomes are assessed by stuff D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- percutaneous stimulation (Experimental): PENS in 2/100HZ, 30 min for each time, twice a day, for 3 days. With conventional analgesic medication if necessary.
  Interventions: Device: PENS
- trancutaneous stimulation (Experimental): TENS in 2/100HZ, 30 min for each time, twice a day, for 3 days. With conventional analgesic medication if necessary.
  Interventions: Device: TENS
- Control (No Intervention): Conventional analgesic medication is offered.

INTERVENTIONS:
Device: PENS — percutaneous electrical nerve stimulation
  Arms: percutaneous stimulation
Device: TENS — transcutaneous electrical nerve stimulation
  Arms: trancutaneous stimulation

SUMMARY:
This study evaluates the effect of percutaneous electrical nerve stimulation (PENS) and transcutaneous nerve stimulation (TENS) for pain relieving in patients with pancreatic cancer. Patients will randomly allocated into PENS group, Tens group and control group.

DETAILED DESCRIPTION:
PENS and TENS have been reported with analgesic effect in patients with pain, including cancer pain, lower back pain, neck pain, stomachache and so on.

Effect and mechanism of PENS on pain relieving has been widely researched. With additional electrical stimulation in certain frequency and intensity to conventional acupuncture, pain controlling effect has been largely enhanced. However, invasive operation limits its application and acceptability, especially on pancreatic cancer.

TENS is an advanced technique generated from PENS, which is much more welcome for its noninvasive character. Further more, its analgesic effect on cancer pain has been proved by several multi-central, randomized, clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic cancer with pain;
* Haven't underwent neurolytic celiac plexus block in the past 1 month;
* With anticipatory survival of more than 3 months.

Exclusion Criteria:

* Metastatic pancreatic cancer;
* Can not tolerate 30 min of lieing in prostrate or side position;
* PS>3;
* Who has been recruited in other clinical trial for pain releiving;
* Who underwent radiotherapy or local radiactive seeds implantation for pain releiving in the past month;
* Imaging diagnosed with encephalic tumor or metastasis;
* Who with cardiac pacemaker or metal stand;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2019-08-26 (Actual)

PRIMARY OUTCOMES:
visal analogue scale (VAS) score | D0-D6
  VAS score before,during and 3 days after treatment

SECONDARY OUTCOMES:
quantity of analgesic medication | D0-D6
  decreasing in quantity of analgesic medication
times of breakthrough pain (BTP) | D0-D6
  times of BTP per day before,during and 3 days after treatment

OTHER OUTCOMES:
complications | D1-D2
  any correlated complications happen during or after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, Dr., Study Chair — Fuda Cancer Hospital
Locations (1):
- Fuda Cancer Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Hurlow A, Bennett MI, Robb KA, Johnson MI, Simpson KH, Oxberry SG. Transcutaneous electric nerve stimulation (TENS) for cancer pain in adults. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD006276. doi: 10.1002/14651858.CD006276.pub3. PMID 22419313
- [Result] Peng L, Min S, Zejun Z, Wei K, Bennett MI. Spinal cord stimulation for cancer-related pain in adults. Cochrane Database Syst Rev. 2015 Jun 29;2015(6):CD009389. doi: 10.1002/14651858.CD009389.pub3. PMID 26121600
- [Result] Chen H, Liu TY, Kuai L, Zhu J, Wu CJ, Liu LM. Electroacupuncture treatment for pancreatic cancer pain: a randomized controlled trial. Pancreatology. 2013 Nov-Dec;13(6):594-7. doi: 10.1016/j.pan.2013.10.007. Epub 2013 Oct 23. PMID 24280575
- [Result] Paley CA, Johnson MI, Tashani OA, Bagnall AM. Acupuncture for cancer pain in adults. Cochrane Database Syst Rev. 2015 Oct 15;2015(10):CD007753. doi: 10.1002/14651858.CD007753.pub3. PMID 26468973
- [Derived] He L, Tan K, Lin X, Yi H, Wang X, Zhang J, Lin J, Lin L. Multicenter, randomized, double-blind, controlled trial of transcutaneous electrical nerve stimulation for pancreatic cancer related pain. Medicine (Baltimore). 2021 Feb 5;100(5):e23748. doi: 10.1097/MD.0000000000023748. PMID 33592831